CLINICAL TRIAL: NCT03068065
Title: Comparison of Efficacy of Liraglutide, Metformin and Gliclazide MR on Hepatic Lipid Content in Patients With Type 2 Diabetes (T2DM) and Non-alcoholic Fatty Liver (NAFLD)
Brief Title: Antidiabetic Effects on Intrahepatic Fat
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Dalong Zhu, Chief physician, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ChiCTR-TRC-14004660
Record Dates: First submitted 2017-02-16; First posted 2017-03-01 (Actual); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Type2 Diabetes
Keywords: Liraglutide; Metformin; Gliclazide
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Liraglutide; Metformin; Gliclazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Liraglutide (Active Comparator): the dosage of liraglutide was 0.6 mg/day during the first week, 1.2 mg/day during the second week, and 1.8 mg/day from the third week to the conclusion of the study
  Interventions: Drug: Liraglutide
- Metformin (Active Comparator): the dosage of merformin was 250 mg thrice a day during the first week, 500 mg thrice a day during the second week, and 1000 mg twice a day from the third week to the conclusion of the study
  Interventions: Drug: Metformin
- Gliclazide (Active Comparator): the initial dosage of gliclazide was 30 mg before breakfast, which was gradually titrated to a maximum of 120 mg/day to achieve a fasting capillary plasma glucose of <7.0 mmol/L
  Interventions: Drug: Gliclazide

INTERVENTIONS:
Drug: Liraglutide — the dosage of liraglutide was 0.6 mg/day during the first week, 1.2 mg/day during the second week, and 1.8 mg/day from the third week to the conclusion of the study
  Other Names: Victoza,Novo Nordisk
  Arms: Liraglutide
Drug: Metformin — the dosage of metformin was 250 mg thrice a day during the first week, 500 mg thrice a day during the second week, and 1000 mg twice a day from the third week to the conclusion of the study
  Other Names: Glucophage,Bristol-Myers Squibb
  Arms: Metformin
Drug: Gliclazide — the initial dosage of gliclazide was 30 mg before breakfast, which was gradually titrated to a maximum of 120 mg/day to achieve a fasting capillary plasma glucose of <7.0 mmol/L
  Other Names: Diamicron MR,Servier
  Arms: Gliclazide

SUMMARY:
This was a 24-week single-center, open-label, parallel controlled group comparing gliclazide, liraglutide, and metformin effects on diabetes with nonalcoholic fatty liver disease.

DETAILED DESCRIPTION:
Following enrollment, eligible participants were randomized (1:1:1) using computer-generated random numbers to the metformin (Glucophage, Bristol-Myers Squibb), liraglutide (Victoza, Novo Nordisk), or gliclazide (Diamicron, Servier) groups. All patients were informed about a proper diet and exercise. For the metformin group (n = 31), the dosage was 250 mg thrice a day during the first week, 500 mg thrice a day during the second week, and 1000 mg twice a day from the third week to the conclusion of the study. For the gliclazide group (n = 31), the initial dosage was 30 mg before breakfast, which was gradually titrated to a maximum of 120 mg/day to achieve a fasting capillary plasma glucose of <7.0 mmol/L. For the liraglutide group (n = 31), the dosage was 0.6 mg/day during the first week, 1.2 mg/day during the second week, and 1.8 mg/day from the third week to the conclusion of the study.At the end of the study, data will be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-70 years;
2. Type 2 diabetes mellitus;
3. Not used antidiabetic drugs within 3 months;
4. HbA1c(7-10%);
5. Presence of fatty liver disease (hepatic fat content ≥ 20% by quantitative ultrasonography);
6. Female subjects：post-menopausal women, take contraceptive measures three months before the test screening and can persist throughout the experimental period;
7. Body mass index (BMI) 20-35kg/m2, and stable Weight 3 months(less than 10% volatility);
8. patients signed the informed consent.

Exclusion Criteria:

1. Used antidiabetic drugs or any other possible hepatic steatosis associated with drugs within the past three months;
2. Suffering from pancreatitis or other pancreatic diseases or have other similar history;
3. GLP-1 analogs or sulfonylurea allergy history;
4. Liver dysfunction (aspartate aminotransferase ≥ 2.5 times of the normalupper limit);
5. Moderate to severe renal insufficiency (eGFR<60ml/min/1.73m2,calculated according to MDRD);
6. Female subjects drinking> 14 units / week; male subjects drinking> 21 units/week;
7. A history of metabolic or autoimmune liver diseases or viral hepatitis diseases;
8. A history of medullary thyroid carcinoma, multiple endocrine neoplasia 2 or family history;
9. Congestive heart failure (NYHA grade Ⅲ - Ⅳ grade);
10. Severe gastrointestinal diseases;
11. Other serious concomitant diseases;
12. Pregnant or planning pregnancy;
13. The researchers believe that the subjects with proliferative retinopathy or macular degeneration need urgentl treatment;
14. Subjects are using unknown ingredients or non herbal medicine preparations or local medicine, researchers believe that during the test the dose of traditional Chinese medicines can not be adjusted or disabled.

Ages: 17 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Intrahepatic fat | -7±3days; 168±3days
  intrahepatic fat change from baseline by quantitative ultrasound

SECONDARY OUTCOMES:
Liver function | -7±3days; 28±3days; 84±3days; 168±3days
  serum alanine aminotransferase (ALT) and serum aspartate aminotransferase (AST)
Lipid | -7±3days; 28±3days; 84±3days; 168±3days
  total cholesterol (CH), triglyceride (TG), high-density lipoprotein cholesterol (HDL), and low-density lipoprotein cholesterol (LDL)
Plasma glucose in standard meal tolerance test | -7±3days; 168±3days
  plasma glucose was measured at 0, 30, 60, and 120 min after ingestion of the meal
Plasma insulin in standard meal tolerance test | -7±3days; 168±3days
  plasma insulin was measured at 0, 30, 60, and 120 min after ingestion of the meal
Glucose control | 14±3days; 28±3days; 56±3days; 84±3days; 112±3days; 140±3days; 168±3days
  fasting blood glucose (FBG), postprandial blood glucose (PBG)
HbA1c | -7±3days; 84±3days; 168±3days
  glycosylated hemoglobin A 1c (HbA1c) was measured by high-performance liquid chromatography
Body composition | -7±3days; 168±3days
  fat mass and lean tissue were measured by dual-energy X-ray absorptiometry
Weight | 14±3days; 28±3days; 56±3days; 84±3days; 112±3days; 140±3days; 168±3days
  body weight
WC | 14±3days; 28±3days; 56±3days; 84±3days; 112±3days; 140±3days; 168±3days
  waist circumference

OTHER OUTCOMES:
Number of Participants with gliclazide, liraglutide or metformin adverse events as a measure of safety and tolerability | -7±3days; 0±3days; 14±3days; 28±3days; 56±3days; 84±3days; 112±3days; 140±3day;168±3days
  adverse events caused by the drugs

CONTACTS AND LOCATIONS:
Overall Officials: Dalong Zhu, MD,PhD, Principal Investigator — the Affiliated Drum Tower Hospital of Nanjing University
Locations (1):
- at Division of Endocrinology, the Affiliated Drum Tower Hospital of Nanjing University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided